CLINICAL TRIAL: NCT02569151
Title: USEFULNESS OF MORNING HOME BLOOD PRESSURE MEASUREMENTS IN JAPANESE PATIENTS WITH TYPE 2 DIABETES MELLITUS: RESULTS OF A 20-YEARS, PROSPECTIVE, LONGITUDINAL STUDY
Brief Title: 20 Years Results by HBP and DBP in Patients With Type 2 Diabetes Mellitus After Following-up
Status: Not yet recruiting | Type: Observational
Sponsor: Kyuzi Kamoi (Other)
Responsible Party: Sponsor-Investigator, Kyuzi Kamoi, eMD & Chief, Nagaoka Red Cross Hospital
Organization: Nagaoka Red Cross Hospital (Other)
Other Study IDs: 9-Kamoi
Record Dates: First submitted 2015-10-05; First posted 2015-10-06 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: HBP & CBP measurement using systo 130 mmHg

SUMMARY:
Participants were examined using the methods reported previous. All chemical laboratory data were obtained at each clinic visit in the morning in a non-fasting state. A single specimen at each visit was used to assess urinary albumin levels based on the 2009 guidelines of the ADA. CBP was measured once in each clinic visit. HBP was measured every day in the morning within 10 minutes after awakening in the sitting position, but HBP value assessed for this study used the value measured once in the same morning at each clinic visit.

Clinic hypertension (CH) and morning hypertension (MH) were defined as systolic BP (SBP) 130 mmHg and/or diastolic BP (DBP) 85 mmHg; clinic normotension (CN) and morning normotension (MN) were defined as SBP <130 mmHg and DBP <85 mmHg, respectively. The reason underlying that same threshold was used for both clinic and morning values was based on criteria of the 1999 WHO-International Society of Hypertension guidelines, because this study started in 1999. Based on HBP, subjects were divided into MH and MN patients, and anti-hypertensive drug use was determined in each group. In addition, based on CBP, subjects were divided into CH and CN patients. These patients were followed using the same methods used for MH and MN patients.

Outcome considered only the first event in each subject. Primary end-point was death from any cause. Secondary end-points were new, worsened, or improved microvascular and macrovascular events.

Risk factors related to each outcome were determined, and therapy which was added to baseline used for each disease in patients with MH was recorded at base- and end-points.

All results are presented as means ± SD. Mean values were compared using the paired or unpaired student t test. To compare the prevalence of events or medical treatment in patients with and without HT on basis of HBP or CBP, Fisher's exact test with two-tailed P values was used, and then hazard ratio and 95% confidence intervals were calculated.

Differences in outcomes between patients with HT and NT on basis of HBP or CBP at base- and end-points in the home or in the clinic, respectively, were assessed using Kaplan-Meier survival curves and then compared by hazard rate using the log-rank test.

Risk factors determined to be statistically related to outcomes were assessed by Cox proportional hazard analysis.

DETAILED DESCRIPTION:
Microalbuminuria and clinical albuminuria were defined as urinary albumin excretion rate 30 mg/g creatinine and 300 mg/g creatinine, respectively (6).

CBP was measured once in each clinic visit. HBP was measured every day in the morning within 10 minutes after awakening in the sitting position, but HBP value assessed for this study used the value measured once in the same morning at each clinic visit.

Clinic hypertension (CH) and morning hypertension (MH) were defined as systolic BP (SBP) 130 mmHg and/or diastolic BP (DBP) 85 mmHg; clinic normotension (CN) and morning normotension (MN) were defined as SBP <130 mmHg and DBP <85 mmHg, respectively. .

Microvascular complications included nephropathy, neuropathy, and retinopathy. Severity of nephropathy was determined based on albuminuria using four categories: normal, 0 points; microalbuminuria, 1 point; clinical albuminuria, 2 points; and dialysis, 3 points. Severity of neuropathy was categorized as normal, 0 points; chronic sensorimotor distal symmetric polyneuropathy and/or cardiac autonomic neuropathy, 1 point. Severity of retinopathy was determined using four categories: normal, 0 points; simple, 1 point; pre-proliferative, 2 points; and proliferative, 3 points. Development of new, worsened, or improved microangiopathy was defined according to a change of at least one step from baseline.

Macrovascular complications included coronary heart disease, cerebrovascular disease and peripheral artery obstruction. Severity of macrovascular events was categorized using two categories: normal, 0 points; and coronary heart disease, cerebrovascular disease, or peripheral artery obstruction, 1 point (3). New, worsened (recurrent), or improved events were defined based on clinical manifestations and treatment throughout the study.

For ethical reasons, patients were treated with various anti-hypertensive, anti-diabetic, anti-dyslipidemia, anti-hypercoagulation and other agents during course of the study by their own doctors.

Outcome results considered only the first event in each subject (3). Primary end-point was death from any cause (3). Secondary end-points were new, worsened, or improved microvascular and macrovascular events (3).

4) Risk factor assessment for outcomes. Risk factors at end-point in ? participants related to each outcome were determined, and therapy which was added to baseline therapy used for each disease in patients with MH was recorded at base- and end-points (3). The 6-month interval minimizes bias due to the fall or rise in the HBP or CBP measurement (10).

Statistical analysis.

1) Baseline. All results are presented as means ± SD. Mean values were compared using the paired or unpaired student t test. To compare the prevalence of micro- and macrovascular complications or medical treatment in patients with and without HT on basis of HBP or CBP (3), Fisher's exact test with two-tailed P values was used, and then hazard ratio and 95% confidence intervals were calculatein.

End-points and outcome measures. Differences in outcomes for each end-point of death, and micro- and macrovascular complications between patients with HT and NT on basis of HBP or CBP at base- and end-points in the home or in the clinic, respectively, were assessed using Kaplan-Meier survival curves and then compared by hazard rate using the log-rank test.

Risk factor assessment for outcomes. Risk factors determined to be statistically related to outcomes were assessed by Cox proportional hazard analysis.

Analysis was performed using the Prism version software (GraphPad Software, CA, USA) and the Statistical Package for the Bioscience (ComWorks Co,Tokyo,Japan). Two-tailed values of P<0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes mellitus

Exclusion Criteria:

* Patients with type 1 diabetes mellitus and with other diseases except diabetes mellitus

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 600 patients with type 2 diabetes mellitus
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-04; Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Death | 20 years

SECONDARY OUTCOMES:
new, worsened, or improved microvascular and macrovascular events | 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Kyuzi Kamoi, MD, Principal Investigator — Jyoetsu General Hospital

REFERENCES:
- [Background] Kamoi K, Miyakoshi M, Soda S, Kaneko S, Nakagawa O. Usefulness of home blood pressure measurement in the morning in type 2 diabetic patients. Diabetes Care. 2002 Dec;25(12):2218-23. doi: 10.2337/diacare.25.12.2218. PMID 12453964
- [Background] Kamoi K. Usefulness of morning home blood pressure measurements in patients with type 2 diabetes mellitus: results of a 10-year, prospective, longitudinal study. Clin Exp Hypertens. 2015;37(2):122-7. doi: 10.3109/10641963.2014.913606. Epub 2014 Apr 30. PMID 24786228